CLINICAL TRIAL: NCT03818048
Title: Inhaled Sevofluran vs Endovenous Propofol for Sedation Maintenance in Patients Submitted to Colonoscopy
Brief Title: Inhaled Sevofluran vs Endovenous Propofol for Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Medico Docente la Trinidad (Other)
Responsible Party: Principal Investigator, Leopoldo Wulff, Principal Investigator, anesthesiologist., Centro Medico Docente la Trinidad
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CMDLT
Record Dates: First submitted 2019-01-04; First posted 2019-01-28 (Actual); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Anesthesia
Keywords: sedation; colonoscopy
MeSH Terms: interventions — Propofol; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group Propofol (Experimental): propofol infusion
  Interventions: Drug: Propofol
- Group Sevoflurane (Experimental): inhalation with sevoflurane
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Propofol — after inicial bolus of propofol, remained sedated with propofol infusion (1-2 mg/kg/min)
  Arms: Group Propofol
Drug: Sevoflurane — after inicial bolus of propofol, remained sedated by inhalation with sevoflurane at a concentration of 2 vol% through a nasal cannula with an oxygen flow.
  Arms: Group Sevoflurane

SUMMARY:
To compare the anesthetic efficacy of the inhalation versus intravenous technique for maintenance of sedation in patients undergoing endoscopy.

A longitudinal, randomized clinical study of 32 patients of both sexes ASA I-III, aged 18-80 years undergoing diagnostic colonoscopy, which was randomly divided into 2 groups. In both, intravenous induction with propofol (2-2.5 mg / kg) was performed, Group A remained sedated with propofol infusion (1-2 mg / kg / min); Group B by inhalation with sevoflurane at a concentration of 2 vol% through a nasal cannula with an oxygen flow.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years
* physical status I, II and III according to the criteria of the American Society of Anesthesiology (ASA)
* patients who are going to undergo diagnostic colonoscopies
* patients who signed the informed consent

Exclusion Criteria:

* Allergy or hypersensitivity to some of the reference drugs in the study
* patients with proven liver disease
* suspicion or confirmation of pregnancy
* antecedent or risk of malignant hyperthermia
* fasting less than 8 hours
* patients with psychic disorders or mental incapacity that make it difficult to understand their participation in the study
* patients who have acute illnesses that compromise their health for which the study cannot be performed

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-10-01 (Actual); Study Completion 2016-12-28 (Actual)

PRIMARY OUTCOMES:
Heart rate | During the colonoscopy - an estimated mean time of 20 minutes
  heart rate per minute
The Recovery Time | 30 min
  Every 5 minutes till a score of 10/10 achieved on Aldrete Score
Propofol dosage | During the colonoscopy - an estimated mean time of 20 minutes
  propofol rescate bolus administered
arterial pressure | During the colonoscopy - an estimated mean time of 20 minutes
  non invasive arterial pressure every 5 minutes
oxygen saturation | During the colonoscopy - an estimated mean time of 20 minutes
  pulse oximetry

SECONDARY OUTCOMES:
adverse reactions in patients | 1 day (postoperative)
  desaturation, laryngospasm
Endoscopist Satisfaction | 60 min
  Endoscopist Satisfaction scored from 1-10. Will be tested on a numerical scale from 0 (not satisfied at all) to 10 (fully satisfied)
Qualitatively assess patient comfort after sedation. | Up to 1 hour after completing the study.
  poor, regular or good

IPD SHARING:
Plan to Share IPD: No